CLINICAL TRIAL: NCT00932997
Title: Reducing the Burden of Breast Cancer Among African American and Latina Survivors
Brief Title: Survivorship Booklets With or Without Individual Telephone Sessions in Increasing Knowledge About the Impact of Breast Cancer in African American and Latina Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 06102; P30CA033572 (NIH); CHNMC-06102; CDR0000642414 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer; Cancer Survivor; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; cancer survivor
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: telephone-based intervention — Participants receive a "Survivorship Kit" and telephone sessions based upon responses to initial survey
Other: counseling intervention — Participants receive a "Survivorship Kit" and telephone sessions based upon responses to initial survey
Other: educational intervention — Participants receive a "Survivorship Kit" alone or in combination with telephone sessions based upon responses to initial survey
Other: questionnaire administration — Baseline and 9 months after enrollment and intervention
Procedure: psychosocial assessment and care — Participants receive a "Survivorship Kit" alone or in combination with telephone sessions based upon responses to initial survey
Procedure: quality-of-life assessment — Baseline and 9 months after enrollment and intervention

SUMMARY:
RATIONALE: Telephone sessions and survivorship booklets may increase knowledge about the psychological and physical impact of breast cancer and increase awareness of available resources. It is not yet known whether survivorship booklets are more effective when given alone or together with individual telephone sessions in informing breast cancer survivors.

PURPOSE: This randomized clinical trial is studying individual telephone sessions given together with survivorship booklets compared with survivorship booklets alone to see how well they work in increasing knowledge about the impact of breast cancer in African American and Latina breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the utility of individual telephone sessions plus survivorship booklets versus the survivorship booklets alone in increasing knowledge about the psychological and physical impact of breast cancer and increasing awareness of appropriate psychological and medical resources among African American and Latina breast cancer survivors.
* Evaluate the utility of these interventions in improving psychological functioning (depression and anxiety) among breast cancer survivors.
* Evaluate the utility of these interventions in improving family and social functioning (changes in family and partner communications) among breast cancer survivors.

Secondary

* Evaluate predictors of health-related quality of life (demographic, medical care factors, psychological, socio-ecological, and socio-cultural factors) within and across breast cancer survivors ethnic groups to identify both general and ethnic-specific correlates.

OUTLINE: Patients are stratified according to ethnicity (African American vs Latina). Patients are randomized to 1 of 2 groups.

* Group 1: Patients receive a survivorship kit of booklets in English or Spanish. Patients then receive a follow-up telephone call at approximately 2 months to clarify any issues relevant to the survivorship kit of booklets.
* Group 2: Patients participate in 8 weekly telephone sessions addressing basic breast cancer information; education about psychological and medical effects of cancer and its treatments; resources including psychosocial, medical care facilities, and clinical trials information; stress management and relaxation; cognitive reframing of concerns and behavioral strategies; family communication; relational communication and intimacy; and social support. Patients also receive a survivorship kit of booklets as in group 1.

After completion of study intervention, patients complete follow-up questionnaires at 4 to 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with breast cancer within the past 1-5 years

  * Stage I-IIIA disease
* No metastatic disease

PATIENT CHARACTERISTICS:

* No other major disabling medical (e.g., another cancer, stroke, heart disease) or psychiatric conditions
* Self-identified ethnically as African-American or Latina
* Able to read and/or speak English or Spanish
* No severe depression or anxiety

  * History of mild to moderate depression or anxiety allowed
* Not pregnant
* Not incarcerated

PRIOR CONCURRENT THERAPY:

* Any type of prior anticancer therapy allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Increased knowledge about the psychological and physical impact of breast cancer | 9 months post study enrollment
Improved psychological functioning (depression and anxiety) | 9 months post study enrollment
Improved family and social functioning (changes in family and partner communications) | 9 months post study enrollment

SECONDARY OUTCOMES:
Predictors of health-related quality of life (demographic, medical care factors, psychological, socio-ecological, and socio-cultural factors) | 9 months post study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kimlin Ashing-Giwa, PhD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States